CLINICAL TRIAL: NCT01890590
Title: A Phase II Study of Cyberknife Radiosurgery for Renal Cell Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Irving Kaplan, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-235
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal Cell Carcinoma; Cyberknife
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Cyberknife treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyberknife (Experimental): You will receive a series of Cyberknife Radiosurgery treatments, with the amount of radiation dosing adjusted for the size of your tumor. The treatment will ideally take place over the course of 3-4 days, but not more than 14 days overall. (3 or 4 fractions of radiation therapy delivered by cyberknife)
  Interventions: Device: CyberKnife

INTERVENTIONS:
Device: CyberKnife — Stereotactic Body Radiation Therapy. 3 or 4 fractions of radiotherapy delivered by Cyberknife.
  Other Names: SBRT

SUMMARY:
CyberKnife Based Radiosurgery is a way to deliver large doses of radiation very accurately to a tumor. The ability of this technology to minimize radiation dose to organs adjacent to the target tumor allows a high dose to be delivered to the tumor, thus potentially increasing the efficacy of radiation treatment. Currently, radiosurgery is commonly used for brain metastases, Stage I lung cancer, spine tumors, and localized prostate cancer. The purpose of this protocol is to evaluate the role of Radiosurgery for the treatment of clinically localized primary renal cell carcinoma.

DETAILED DESCRIPTION:
Before the research starts (screening) Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about your health, current medications, and any allergies.
* Performance status, which evaluates how you are able to carry on with your usual activities.
* Quality of life survey.
* Gold seed (Fiducial) Placement: Placement of at least one (usually up to 3) gold fiducial(s) must be placed in or around the tumor by a surgeon or interventional radiologist a minimum of one week or more prior to pre-treatment planning simulation.
* An assessment of your tumor by X-ray, CT (Computerized Tomography) scan, MRI (Magnetic Resonance Imaging) or PET (Positron Emission Tomography) scans.
* Blood tests.
* Urine test.
* You will undergo a simulation of the intervention procedure. It will involve the study team helping you position yourself for the study procedure as you undergo a CT scan of the abdomen while holding the correct position.

If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

After the screening procedures confirm that you are eligible to participate in the research study:

You will receive a series of Cyberknife Radiosurgery treatments, with the amount of radiation dosing adjusted for the size of your tumor. The treatment will ideally take place over the course of 3-4 days, but not more than 14 days overall.

You will be positioned in a stable position laying on your back, capable for reproducibility of positioning and not allowing you to move from simulation to treatment, allowing you to feel as comfortable as possible. A variety of systems may be utilized to keep you still; including vacuum bag, alpha cradle, or stereotactic frames that surround you on three sides and large rigid pillows conforming to your body.

After the final dosing We would like to keep track of your medical condition for the rest of your life. We would like to do this by calling you on the telephone once a year to see how you are doing. Keeping in touch with you and checking your condition every year helps us look at the long-term effects of the research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically or radiological evidence of Stage I (T1N0M0) renal cell carcinoma with a size no larger than 8 cm in greatest dimension measured by MRI or CT Scan
* At least one (usually up to 3) gold fiducial placed in or around tumor, can be performed on the same day - after signing research informed consent.
* No irreversible coagulopathies
* Age ≥ 18 years old because no dosing or adverse event data are currently available on the use of Cyberknife Radiosurgery radiation in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric Phase II trials.
* ECOG Performance Status ≤2 (Appendix A).
* At least 12 month life expectancy
* Ability to have CT and/or MRI imaging with or without contrast and must be performed within 120 days prior to registration.
* No other cancer in previous 2 years with the exception of non-invasive skin cancers
* All subjects meeting eligibility criteria irrespective of gender, minority or other underrepresented status will be eligible for enrollment into the study.
* The effects of Cyberknife Radiosurgery on the developing human fetus are unknown. For this reason and because Radiation is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document and study specific consent form prior to study entry.
* Labs: Serum Creatinin <3 mg/dl, Urinalysis, INR <2, PTT <70 sec, AST, ALT ≤2.5x ULN, Abnormalities on urinalysis (i.e. proteinuria) will not exclude patients from participation on study.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Irreversible coagulopathies that preclude fiducial placement
* Prior upper abdominal external beam irradiation
* Prior history of invasive malignancy within the last 2 years
* Inability to deliver target dose with CyberKnife due to inability to image fiducials
* Inability to deliver target dose with CyberKnife due to normal tissue dose constraints
* Inability to have contrast CT or MRI to help define tumor volume for radiation planning
* Decreased platelet count and / or anticoagulation parameters that would preclude transcutaneous placement of fiducials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
To determine the freedom from local tumor progression in patients treated with CyberKnife radiosurgery for primary renal tumors at 6 months | 2 Years
  To determine the freedom from local tumor progression in patients treated with CyberKnife radiosurgery for primary renal tumors at 6 months

SECONDARY OUTCOMES:
To determine impact of therapy on quality of life. | 2 Years
  To determine impact of therapy on quality of life.
To evaluate adverse events. | 2 years
  To evaluate adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Irving D Kaplan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No